CLINICAL TRIAL: NCT04042532
Title: The Effects and Mechanisms of Theta-burst Stimulation on Cognitive Function in the Patients with Biomarker-defined Young-onset Alzheimer's Disease Dementia
Brief Title: Theta-burst Stimulation on Cognitive Function in the Patients with Young-onset Alzheimer's Disease Dementia
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 201802104A0
Record Dates: First submitted 2019-07-28; First posted 2019-08-02 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Alzheimer Disease, Early Onset
Keywords: Young-onset dementia; Alzheimer's disease; rTMS; TBS
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Active group (Active Comparator): Active group will receive active stimulation of standard intermittent TBS (iTBS) protocol.
  Interventions: Device: Theta-burst stimulation (TBS)
- Sham group (Sham Comparator): Sham group will receive sham stimulation of the same iTBS protocol with the coil set at 90 to the skull.
  Interventions: Device: Theta-burst stimulation (TBS)
- Cognitively normal control (No Intervention): Cognitively normal controls will be recruited for neuroimaging comparison.

INTERVENTIONS:
Device: Theta-burst stimulation (TBS) — We will perform standard intermittent TBS (iTBS) parameters to left DLPFC of every patient in the study. The frequency parameters of TBS are 3-pulse 50-Hz bursts, every 200 ms at 5 Hz, and the intensity is 90% of active motor threshold. A single session of iTBS contains 2 s of TBS repeated every 10 s for 20 times. In this study, we will give two sessions of iTBS separated by 15 min.
  Arms: Active group; Sham group

SUMMARY:
Young-onset dementia (YOD) is a devastating condition, and it produces substantial psychosocial impacts on individual's functioning and family's care burden. Alzheimer's disease (AD) dementia is the most common type in YOD. Medication treatment Response was limited and unsatisfactory. In recent years, repetitive transcranial magnetic stimulation (rTMS) has been considered an alternative for the improvement of cognition in older patients with cognitive impairment. This study aims to examine the effects and potential mechanisms of theta-burst stimulation (TBS) on cognitive function in individuals with young-onset AD.

DETAILED DESCRIPTION:
The investigators apply the National Institute on Aging-Alzheimer's Association (NIA-AA) criteria to recruit the biomarker-defined, young-onset AD patients with intermediate-to-high levels of biological evidence. This is a randomized, sham-controlled, 2-way crossover study, and combined neuroimaging study of 18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose (18F-FDG) positron emission tomography (PET) to further explore the potential mechanisms. This study will consist of two intervention periods. A total of 50 young-onset AD patients will be consecutively recruited and be randomized into one of two groups: active and sham stimulation (n = 25 per group) in every intervention period. Besides, 20 cognitively normal subjects will be recruited for neuroimaging comparison. Cognitive evaluation will be performed before and immediately after treatment at 2 weeks of TBS intervention, and 4 weeks after TBS. Data on functional neuroimaging will be also collected before and after TBS protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Any patient has a definite diagnosis of AD dementia according to the NIA-AA criteria for intermediate-to-high levels of biological evidence of probable and possible AD dementia (McKhann et al. 2011).
2. Dementia onset before age 65 years old.
3. Age between 50-75 years old for patient and control group.
4. The severity of dementia is limited to mild to moderate stage in current project. The definition of mild to moderate stage of dementia is based on the clinical dementia rating scale (CDR) from 0.5-2.
5. Cognitively normal controls MMSE≧24, CDR should be 0.
6. Informed consent provided by the patient and family.

Exclusion Criteria:

1. Any subject has a definite diagnosis of epilepsy or history of seizure attack.
2. Current or past history of clinically significant neurological insults affecting brain structure or function like completed stroke, head injury or brain tumor.
3. Any subject has clinically significant or unstable medical diseases including metabolic, renal, liver, lung or cardiovascular disorders including metabolic, renal, liver, lung or cardiovascular disorders
4. Any subject has current alcohol or other substances abuse and/ or dependence within the recent one year, or previously prolonged history of substances abuse
5. Any females who is pregnant or lactating
6. General MRI, TMS and/or PET exclusion criteria including subjects who had received brain aneurysm surgery, or implanted pacemaker, mechanical valves, cochlear implant or other metal devices/ objects that are not magnetic resonance (MR) compatible in the body.
7. Any subject has allergic reaction to 18F-florbetapir or 18F-FDG radiotracers.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-01-03 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline MMSE total scores immediately after TBS intervention | Before and immediately after TBS intervention
  The changes of Mini-Mental State Examination (MMSE) total scores (score range from 0 to 30, higher values represent a better cognitive outcome)
Change from baseline MMSE total scores 4 weeks after TBS intervention | Before and 4 weeks after TBS intervention
  The changes of Mini-Mental State Examination (MMSE) total scores (score range from 0 to 30, higher values represent a better cognitive outcome)
Change from baseline ADAS-Cog total scores immediately after TBS intervention | Before and immediately after TBS intervention
  The changes of Alzheimer's Disease Assessment Scale-Cognitive (ADAS-Cog) total scores (score range from 0 to 70, higher score indicates a worse cognitive outcome)
Change from baseline ADAS-Cog total scores 4 weeks after TBS intervention | Before and 4 weeks after TBS intervention
  The changes of Alzheimer's Disease Assessment Scale-Cognitive (ADAS-Cog) total scores (score range from 0 to 70, higher score indicates a worse cognitive outcome)

SECONDARY OUTCOMES:
The standard uptake values changes of FDG-PET | Before and 1 week after TBS intervention
  The standard uptake values (SUV) changes of cerebral glucose metabolism using 18F-FDG-PET

CONTACTS AND LOCATIONS:
Overall Officials: KUAN YI WU, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Guishan, Taiwan

IPD SHARING:
Plan to Share IPD: No